CLINICAL TRIAL: NCT02538822
Title: Assessment of the Risk of Rupture of Aneurysms of the Thoracic Ascending Aorta (ATA) From the Dynamic Imaging - A Monocentric Study
Brief Title: Risk of Rupture of Aneurysms of the Thoracic Ascending Aorta (ATA) From the Dynamic Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low inclusion rates
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1408061; ANSM (Other: 2014-A00568-39)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2020-01

CONDITIONS: Aortic Aneurysm, Thoracic
Keywords: aortic aneurysm; thoracic ascending aorta; ATA; dynamic imaging; mechanical testing
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Aneurysm | interventions — Mechanical Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thoracic ascending aorta (ATA) (Experimental): the risk of rupture of thoracic ascending aorta (ATA) is assessed fom the dynamic imaging and mechanical testing
  Interventions: Device: dynamic imaging; Device: mechanical testing

INTERVENTIONS:
Device: dynamic imaging — In vivo study of biomechanical behavior of ATA from preoperative dynamic imaging : dynamic CT-scan and 4D-magnetic resonance imaging (MRI)
Device: mechanical testing — In vitro study of with mechanical inflation testing of ATA tissue harvested during surgery.

SUMMARY:
Aneurysms of the thoracic ascending aorta are a serious pathology which may threatens life by rupture or dissection. Their incidence is estimated at 10.4 per 100,000 people. At present, the only parameter for assessing the risk of complication is the maximum diameter of the aneurysm. The only way to avoid a complication is a surgical replacement of the aneurysmal aorta by a prosthetic tube. This procedure is performed by sternotomy and with extracorporeal circulation and its death rate ranges between 3% and 5%. Surgical repair is indicated when the diameter of the aneurysm exceeds 5.5 cm for degenerative atheromatous aneurysms or 5 cm in a patient with genetic disorder of connective tissue (Marfan disease or Ehlers-Danlos syndrome). However, there are aneurysms with diameter greater than the surgical threshold which remain stable. Conversely, complications have been described for aneurysms less than 4.5 cm in diameter. The criterion of diameter appears therefore as inadequate to assess the risk of complication of an aneurysm of the ascending aorta.Multiple methods have been described in the literature. One of them relies on in vitro mechanical testing on healthy or aneurysmal tissue. Another method is the vivo analysis from imaging (CT, MRI or ultrasound). So far, no algorithm is robust enough for predicting the risk of complication better than the universally used criterion of diameter.

The pathophysiology of these aneurysms has also been explored from histological studies. The investigators know that the microstructure of the aortic wall of an aneurysm is deteriorated with a degradation of elastin fibers and collagen that determine to a large extent its biomechanical behavior. Histological analysis appears inseparable from biomechanical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diameter of ATA exceeds 5.5 cm
* Diameter of ATA exceeds 5 cm in a patient with genetic disorder of connective tissue (Marfan disease or Ehlers-Danlos syndrome)
* Diameter of ATA exceeds 5 cm in a patient with aortic valvulopathy
* Written consent

Exclusion Criteria:

* Contra-indication to MRI
* Chronic insufficiency kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2018-09-16 (Actual); Study Completion 2018-09-16 (Actual)

PRIMARY OUTCOMES:
Correlation between index of risk of the rupture and in vivo physiological elasticity. | day 1
  The index of risk of rupture is a composite measure :
  * an in vivo study of biomechanical behavior of aneurysmal aorta from preoperative dynamic imaging (dynamic CT-scan and 4D-MRI). It will determine the maximum stress borne by the aortic wall and its physiological elasticity.
  * an in vitro study with mechanical inflation testing of aneurysmal aortic tissue harvested during surgery. These tests will be conducted up to rupture and will bring results on the elasticity of the aortic wall of the aneurysm and its mode of failure.
  * finally, a histological analysis, with measurement of elastin and collagen content.
  The physiological elasticity is measured from MRI

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore CAMPISI, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No